CLINICAL TRIAL: NCT01526174
Title: Safety and Efficacy of Intratympanically Delivered Golimumab for Stabilization of Hearing in Patients With Autoimmune Inner Ear Disease: An Open-label Proof-of-concept Clinical Trial
Brief Title: Intratympanic Injection for Autoimmune Inner Ear Disease
Acronym: AIED
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: House Research no longer conducting research.
Sponsor: House Research Institute (Other)
Collaborators: Janssen Services, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRI-002; TNFalpha (Other: House Research Institute)
Record Dates: First submitted 2012-02-01; First posted 2012-02-03 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: Autoimmune Inner Ear Disease
Keywords: autoimmune; hearing loss; bilateral hearing loss; steroid-dependent
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Bilateral | interventions — golimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- First Arm (Experimental): Determine safety of intratympanic injection
  Interventions: Drug: Golimumab
- Second Arm (Experimental): Efficacy evaluation of 4 intratympanic injections
  Interventions: Drug: Golimumab

INTERVENTIONS:
Drug: Golimumab — Intratympanic injection 0.3ml First Arm: 1 injection Second Arm: 4 injections
  Other Names: Simponi

SUMMARY:
The investigators plan to conduct an open-label intratympanic injection proof-of-concept trial of golimumab, a TNF-alpha inhibitor, assessing for hearing loss progression in patients with autoimmune inner ear disease (AIED). This specific aim will be achieved using a two-arm approach. First, the investigators propose to dose 3 individual subjects with a single intratympanic injection of golimumab and follow each for 30 days, closely examining them for adverse events. If there are no serious adverse events, with FDA approval, the investigators propose to dose 14 subjects, each with 4 intratympanic injections of golimumab.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autoimmune inner ear disease (AIED) by the principal investigator
* Idiopathic, bilateral sensorineural hearing loss
* History of, or audiograms showing, rapid progression of hearing loss
* Bilateral loss of at least 30 dB in one or more frequencies (0.25 - 6 kHz)
* Hearing responsive on high-dose oral steroids and steroid-dependent, as determined by history and the principal investigator. The subject can be taking oral steroid, at the maintenance level, if enrolled in the First Arm and, if enrolled in the Second Arm, will begin taper after the first injection.
* Provided written informed consent for participation in the clinical study

Exclusion Criteria:

* Positive MRI for vestibular schwannoma
* Positive FTA (syphilis)
* Significant middle ear disease (e.g., otitis media)
* Positive blood test for Lyme disease
* Positive tuberculosis test
* Concurrent or past treatment or use of medications and/or substances known to cause ototoxicity(for example, aminoglycosides [e.g., gentamicin], cisplatin, loop diuretics, Yorgason et al., 2006)
* Known adverse reaction to golimumab, adalimumab, etanercept, infliximab, rituximab, ustekinumab, or other biologic immunomodulators
* Concurrent (within the past 3 months prior to enrollment) live viral intranasal vaccine (flu)
* Positive test for HIV
* Positive test for Hepatitis B and C
* Presence of a demyelinating disease, such as multiple sclerosis
* Women of childbearing potential only: Positive serum pregnancy test prior to the only/first injection
* Active infections

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-03; Primary Completion 2013-12 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Serious Adverse Events | 30 days
  Serious Adverse Events
Pure-tone threshold change | 6 weeks
  Change in pure-tone threshold from baseline to 6 week after initiation of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Derebery, MD, Principal Investigator — House Research Institute